CLINICAL TRIAL: NCT03572244
Title: Comparison of Pro-Inflammatory Cytokines and Bone Metabolism Mediators Around Laser-Lok and Machined Transmucosal Abutments: A Pilot, Randomized Clinical Trial
Brief Title: Comparing Pro-Inflammatory Cytokines and Bone Metabolism Mediators Around Laser-Lok and Machined Transmucosal Abutments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Barwacz (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Christopher Barwacz, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201507837
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Dental Implants
Keywords: Laser-Lok; Crevicular fluid; Machined; Abutment

STUDY DESIGN:
Intervention Model Description: 6 subjects will be randomized to Laser-Lok placement, and 6 subjects will be randomized to machined healing abutment placement. The assignment will be a 1:1 scheme, with the study coordinator randomly opening pre-assigned envelopes to determine implant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Laser-Lok (Experimental): A Laser-Lok microgrooved implant will be placed.
  Interventions: Device: Laser-Lok
- Machine (Active Comparator): A machined implant will be placed.
  Interventions: Device: Machined

INTERVENTIONS:
Device: Laser-Lok — A microgrooved abutment will be placed
  Arms: Laser-Lok
Device: Machined — A machined transmucosal healing abutment will be placed
  Arms: Machine

SUMMARY:
A pilot, prospective, randomized clinical trial is proposed. It is primarily aimed at assessing the expression of pro-inflammatory cytokine and bone metabolism mediators adjacent to Laser-Lok microgrooved (LL) or machined (M) transmucosal healing abutments. The pilot study would seek recruitment of 12 subjects requiring replacement of a single, toothbound molar or premolar in the maxilla or mandible with an implant-supported restoration.

DETAILED DESCRIPTION:
The purpose of this research study is to compare two different implant abutment designs, microgrooved and machined. The implant abutment is the dental prosthetic part that connects the implant to the crown. As a part of this study, subjects will have a dental implant surgically placed in their jaw bone. The implant will serve as the artificial root. After the implant heals, subjects will have the abutment and crown placed on the implant.

This study will compare levels of inflammation next to the implant abutment. Both implant abutment designs are FDA approved but differ in microtexturing. This study will determine if these texture differences have any impact on the healing of subjects' jaw bone and gums after implant surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Subjects requiring the replacement of either a tooth-bound molar or premolar in either arch that do not require simultaneous implant site development (i.e., bone and/or soft-tissue grafting)
* Teeth adjacent (mesial and distal) to study site must consist of two stable, natural teeth without signs of periodontal attachment loss up to 2.0mm
* An opposing dentition with teeth, implants, or fixed prosthesis
* Subjects must be willing to forgo use of a provisional appliance (e.g., removable interim partial denture (or) "flipper", essix appliance, etc.) during the active portion (from implant placement to 8 week +IP visit) of the study protocol.
* Subjects must be willing to follow instructions related to the study procedures
* Subjects must have read, understood, and signed the informed consent document

Exclusion Criteria:

* Insufficient interocclusal space for implant placement and/or restoration at study site
* Insufficient lateral ridge volume for implant placement in a prosthetically-driven location
* More than 2.0 mm of vertical bone loss at study site as measured from the interproximal crestal bone on the adjacent teeth
* Untreated rampant caries
* Tobacco use free for ≤ 6 months
* Liver or kidney dysfunction/failure
* Active severe infectious diseases that may affect normal healing and/or bone metabolism
* Uncontrolled diabetes determined as HbA1c value > 7%
* Current alcohol or drug abuse
* Need for systemic medications (e.g., corticosteroids) that may influence postoperative healing and/or osseointegration
* History of relevant head/neck cancer and/or radiation of the head/neck within the last 24 months
* Subjects who currently use IV bisphosphonates or have a history of IV bisphosphonate use
* Subjects with metabolic bone diseases such as severe osteoporosis or Paget's disease of bone
* Known pregnancy or nursing mothers
* Unwilling to forgo use of a provisional appliance (e.g., removable interim partial denture (or) "flipper", essix appliance, etc.) during the active portion (from implant placement to 8 week +IP visit) of the study protocol.
* Unable or unwilling to return for follow-up visits for a period of 1 year
* Unlikely to be able to comply with study procedures according to investigators judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Barwacz, DDS, Principal Investigator — The University of Iowa College of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nevins M, Nevins ML, Camelo M, Boyesen JL, Kim DM. Human histologic evidence of a connective tissue attachment to a dental implant. Int J Periodontics Restorative Dent. 2008 Apr;28(2):111-21. PMID 18546807
- [Background] Pecora GE, Ceccarelli R, Bonelli M, Alexander H, Ricci JL. Clinical evaluation of laser microtexturing for soft tissue and bone attachment to dental implants. Implant Dent. 2009 Feb;18(1):57-66. doi: 10.1097/ID.0b013e31818c5a6d. PMID 19212238
- [Background] Shapoff CA, Lahey B, Wasserlauf PA, Kim DM. Radiographic analysis of crestal bone levels around Laser-Lok collar dental implants. Int J Periodontics Restorative Dent. 2010 Apr;30(2):129-37. PMID 20228972
- [Background] Botos S, Yousef H, Zweig B, Flinton R, Weiner S. The effects of laser microtexturing of the dental implant collar on crestal bone levels and peri-implant health. Int J Oral Maxillofac Implants. 2011 May-Jun;26(3):492-8. PMID 21691595
- [Background] Geurs NC, Geisinger ML, Vassilopoulos PJ, O'Neal SJ, Haigh SJ, Reddy MS. Optimizing Connective Tissue Integration on Laser-Ablated Implant Abutments. Clin Adv Periodontics. 2016 Aug;6(3):153-159. doi: 10.1902/cap.2016.150068. PMID 31535464
- [Background] Nevins M, Camelo M, Nevins ML, Schupbach P, Kim DM. Connective tissue attachment to laser-microgrooved abutments: a human histologic case report. Int J Periodontics Restorative Dent. 2012 Aug;32(4):385-92. PMID 22577643
- [Background] Nevins M, Nevins M, Gobbato L, Lee HJ, Wang CW, Kim DM. Maintaining interimplant crestal bone height via a combined platform-switched, Laser-Lok implant/abutment system: a proof-of-principle canine study. Int J Periodontics Restorative Dent. 2013 May-Jun;33(3):261-7. doi: 10.11607/prd.1773. PMID 23593619
- [Background] Norton MR. Understanding the intimate relationship between biomechanics and optimal clinical performance: application of implant design. Compend Contin Educ Dent. 2002 Sep;23(9 Suppl 2):21-5. PMID 12790010
- [Background] Steigenga JT, al-Shammari KF, Nociti FH, Misch CE, Wang HL. Dental implant design and its relationship to long-term implant success. Implant Dent. 2003;12(4):306-17. doi: 10.1097/01.id.0000091140.76130.a1. PMID 14752967
- [Background] Stanford CM. Biomechanical and functional behavior of implants. Adv Dent Res. 1999 Jun;13:88-92. doi: 10.1177/08959374990130012101. PMID 11276753
- [Background] Ratner BD. Replacing and renewing: synthetic materials, biomimetics, and tissue engineering in implant dentistry. J Dent Educ. 2001 Dec;65(12):1340-7. PMID 11780652
- [Background] Lowney JJ, Norton LA, Shafer DM, Rossomando EF. Orthodontic forces increase tumor necrosis factor alpha in the human gingival sulcus. Am J Orthod Dentofacial Orthop. 1995 Nov;108(5):519-24. doi: 10.1016/s0889-5406(95)70052-8. PMID 7484971
- [Background] Fiorellini JP, Nevins ML, Sekler J, Chung A, Oringer RJ. Correlation of peri-implant health and aspartate aminotransferase levels: a cross-sectional clinical study. Int J Oral Maxillofac Implants. 2000 Jul-Aug;15(4):500-4. PMID 10960982
- [Background] Nowzari H, Botero JE, DeGiacomo M, Villacres MC, Rich SK. Microbiology and cytokine levels around healthy dental implants and teeth. Clin Implant Dent Relat Res. 2008 Sep;10(3):166-73. doi: 10.1111/j.1708-8208.2007.00076.x. Epub 2008 Jan 24. PMID 18218050
- [Background] Nowzari H, Phamduong S, Botero JE, Villacres MC, Rich SK. The profile of inflammatory cytokines in gingival crevicular fluid around healthy osseointegrated implants. Clin Implant Dent Relat Res. 2012 Aug;14(4):546-52. doi: 10.1111/j.1708-8208.2010.00299.x. Epub 2010 Jul 17. PMID 20662860
- [Background] Schierano G, Pejrone G, Brusco P, Trombetta A, Martinasso G, Preti G, Canuto RA. TNF-alpha TGF-beta2 and IL-1beta levels in gingival and peri-implant crevicular fluid before and after de novo plaque accumulation. J Clin Periodontol. 2008 Jun;35(6):532-8. doi: 10.1111/j.1600-051X.2008.01224.x. Epub 2008 Apr 1. PMID 18384390
- [Background] Salvi GE, Aglietta M, Eick S, Sculean A, Lang NP, Ramseier CA. Reversibility of experimental peri-implant mucositis compared with experimental gingivitis in humans. Clin Oral Implants Res. 2012 Feb;23(2):182-190. doi: 10.1111/j.1600-0501.2011.02220.x. Epub 2011 Aug 2. PMID 21806683
- [Background] Petkovic AB, Matic SM, Stamatovic NV, Vojvodic DV, Todorovic TM, Lazic ZR, Kozomara RJ. Proinflammatory cytokines (IL-1beta and TNF-alpha) and chemokines (IL-8 and MIP-1alpha) as markers of peri-implant tissue condition. Int J Oral Maxillofac Surg. 2010 May;39(5):478-85. doi: 10.1016/j.ijom.2010.01.014. Epub 2010 Mar 5. PMID 20207110
- [Background] Murata M, Tatsumi J, Kato Y, Suda S, Nunokawa Y, Kobayashi Y, Takeda H, Araki H, Shin K, Okuda K, Miyata T, Yoshie H. Osteocalcin, deoxypyridinoline and interleukin-1beta in peri-implant crevicular fluid of patients with peri-implantitis. Clin Oral Implants Res. 2002 Dec;13(6):637-43. doi: 10.1034/j.1600-0501.2002.130610.x. PMID 12519339
- [Background] Severino VO, Napimoga MH, de Lima Pereira SA. Expression of IL-6, IL-10, IL-17 and IL-8 in the peri-implant crevicular fluid of patients with peri-implantitis. Arch Oral Biol. 2011 Aug;56(8):823-8. doi: 10.1016/j.archoralbio.2011.01.006. Epub 2011 Feb 8. PMID 21306703
- [Background] Javed F, Al-Hezaimi K, Salameh Z, Almas K, Romanos GE. Proinflammatory cytokines in the crevicular fluid of patients with peri-implantitis. Cytokine. 2011 Jan;53(1):8-12. doi: 10.1016/j.cyto.2010.08.013. Epub 2010 Sep 25. PMID 20870421
- [Background] Lachmann S, Kimmerle-Muller E, Axmann D, Scheideler L, Weber H, Haas R. Associations between peri-implant crevicular fluid volume, concentrations of crevicular inflammatory mediators, and composite IL-1A -889 and IL-1B +3954 genotype. A cross-sectional study on implant recall patients with and without clinical signs of peri-implantitis. Clin Oral Implants Res. 2007 Apr;18(2):212-23. doi: 10.1111/j.1600-0501.2006.01322.x. PMID 17348886
- [Background] Andreiotelli M, Koutayas SO, Madianos PN, Strub JR. Relationship between interleukin-1 genotype and peri-implantitis: a literature review. Quintessence Int. 2008 Apr;39(4):289-98. PMID 19081897
- [Background] Boynuegri AD, Yalim M, Nemli SK, Erguder BI, Gokalp P. Effect of different localizations of microgap on clinical parameters and inflammatory cytokines in peri-implant crevicular fluid: a prospective comparative study. Clin Oral Investig. 2012 Apr;16(2):353-61. doi: 10.1007/s00784-010-0497-4. Epub 2011 Jan 7. PMID 21212999
- [Background] Ataoglu H, Alptekin NO, Haliloglu S, Gursel M, Ataoglu T, Serpek B, Durmus E. Interleukin-1beta, tumor necrosis factor-alpha levels and neutrophil elastase activity in peri-implant crevicular fluid. Clin Oral Implants Res. 2002 Oct;13(5):470-6. doi: 10.1034/j.1600-0501.2002.130505.x. PMID 12453123
- [Background] Barwacz CA, Brogden KA, Stanford CM, Dawson DV, Recker EN, Blanchette D. Comparison of pro-inflammatory cytokines and bone metabolism mediators around titanium and zirconia dental implant abutments following a minimum of 6 months of clinical function. Clin Oral Implants Res. 2015 Apr;26(4):e35-e41. doi: 10.1111/clr.12326. Epub 2014 Jan 13. PMID 24417614

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 23 enrolled participants, 12 met the inclusion criteria, were randomized to treatment, and completed the study.
Period: Overall Study
Arm/Group | Laser-Lok | Machine
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser-Lok | Machine | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 62 [52 to 72] | 61 [36 to 79] | 62 [36 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 3 | 1 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Difference in PICF Cytokine Levels (Log pg/ml) for Various Biomarkers, Specifically at Laser-Lok Abutment Sites and Machined Abutment Sites at 8 Weeks After Implant Placement
Description: Determine if there is a difference in peri-implant crevicular fluid's pro-inflammatory and bone-metabolism mediator profiles, specifically for peri-implant crevicular fluid that is next to Laser-Lok microgrooved (LL) and machined (M) healing abutments after a healing period of 8 weeks after implant placement.
Time Frame: 8 weeks after implant placement
Measure: Mean (Standard Deviation); unit: log pg/ml
Arm/Group | Laser-Lok | Machine
Number analyzed (Participants) | 6 | 6
log pg/ml
  logTNFa | 2.25 (1.18) | 2.15 (1.00)
  logIL6 | 1.80 (0.31) | 1.61 (0.36)
  logIL8 | 6.54 (0.60) | 5.52 (1.06)
  logMMP1 | 4.48 (0.64) | 3.89 (0.72)
  logIP10 | 1.29 (0.79) | 1.32 (1.09)
  logMMP8b | 11.37 (0.37) | 10.61 (1.11)
  logIL_1B | 5.19 (0.61) | 4.92 (1.08)
  logMMP13 | 5.73 (0.94) | 5.78 (1.08)
  logENA78 | 4.05 (0.53) | 3.27 (0.65)
  logMIG | 6.95 (0.12) | 6.63 (0.51)
  logOsteopontin | 6.44 (1.19) | 6.50 (0.96)
  logITAC1 | 2.53 (0.36) | 2.56 (0.84)
  logOsteoprotegerin | 2.94 (0.95) | 3.38 (1.06)

2. Primary Outcome: Difference in GCF Cytokine Levels (Log pg/ml) for Various Biomarkers, Specifically at Laser-Lok Abutment Sites and Machined Abutment Sites at 8 Weeks After Implant Placement
Description: Determine if there is a difference in gingival crevicular fluid's pro-inflammatory and bone-metabolism mediator profiles, specifically for gingival crevicular fluid that is next to Laser-Lok microgrooved abutments (LL) and machined (M) habutments after a healing period of 8 weeks after implant placement.
Time Frame: 8 weeks after implant placement
Measure: Mean (Standard Deviation); unit: log pg/ml
Arm/Group | Laser-Lok | Machine
Number analyzed (Participants) | 6 | 6
log pg/ml
  logTNFa | 2.52 (0.50) | 2.13 (1.15)
  logIL6 | 1.86 (0.09) | 2.39 (1.06)
  logIL8 | 6.30 (0.84) | 6.29 (1.31)
  logMMP1 | 4.12 (0.35) | 4.47 (0.62)
  logIP10 | 1.13 (0.84) | 2.05 (2.14)
  logMMP8b | 11.10 (0.50) | 11.17 (0.76)
  logIL_1B | 4.70 (0.82) | 5.06 (0.80)
  logMMP13 | 5.63 (0.36) | 5.18 (1.87)
  logENA78 | 3.94 (0.79) | 3.75 (0.68)
  logMIG | 6.88 (0.18) | 6.95 (0.32)
  logOsteopontin | 6.82 (0.49) | 6.56 (1.21)
  logITAC1 | 2.48 (0.20) | 2.18 (1.01)
  logOsteoprotegerin | 2.84 (1.56) | 3.69 (0.82)

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Laser-Lok | Machine
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
One of the primary limitations is the small sample size (n=12).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-01-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT03572244/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03572244/SAP_001.pdf